CLINICAL TRIAL: NCT03907176
Title: A Phase 3b, Randomized, Open-Label Study of HTX-011 as the Foundation of a Non-opioid, Multimodal Analgesic Regimen to Decrease Opioid Use Following Unilateral Open Inguinal Herniorrhaphy
Brief Title: Herniorrhaphy Study for Opioid Elimination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTX-011-304
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Analgesia
Keywords: inguinal hernia; hernia; hernia surgery; postoperative pain; herniorrhaphy; multimodal analgesia
MeSH Terms: conditions — Agnosia; Hernia, Inguinal; Hernia; Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: In Part 1, subjects who meet the Screening eligibility criteria (Section 4.1) will be randomized to one of the 2 parallel cohorts. In Part 2, prior to surgery, the Investigator will select for the subject one of the 2 postoperative MMA regimens, based on Investigator and/or subject preference.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1 (Experimental): HTX-011; Ibuprofen and Acetaminophen (regimen 1)
  Interventions: Drug: HTX-011; Device: Luer lock applicator; Drug: Ibuprofen; Drug: Acetaminophen
- Cohort 2 (Experimental): HTX-011; Ibuprofen and Acetaminophen (regimen 2)
  Interventions: Drug: HTX-011; Device: Luer lock applicator; Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: HTX-011 — 300 mg
Device: Luer lock applicator — Applicator for instillation
Drug: Ibuprofen — 600 mg
Drug: Acetaminophen — 1 g

SUMMARY:
This is a Phase 3b, open-label study to assess postoperative opioid use in subjects undergoing unilateral open inguinal herniorrhaphy with intraoperative administration of HTX-011 and a postoperative non-opioid multimodal analgesic (MMA) regimen. The study will be conducted in 2 sequential parts: Part 1 is randomized and Part 2 is Investigator's preference for MMA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled and medically fit to undergo an elective unilateral open inguinal herniorrhaphy with mesh under deep sedation or general anesthesia; no neuraxial technique (eg, no spinal or epidural).
* Has an American Society of Anesthesiologists (ASA) Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a planned concurrent surgical procedure (eg, bilateral herniorrhaphy).
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Part 1 only: Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months. Part 2 only: Has known or suspected history of persistent opioid use, defined as daily, or almost daily, use of opioids for a period of at least 30 days within the previous 6 months.
* Has taken any opioids within 24 hours prior to the scheduled surgery.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Has a known or suspected history of drug abuse, has a positive drug screen on the day of surgery, consumes 3 or more alcoholic drinks every day, or has a recent history of alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who do not receive an opioid prescription at discharge through the day 15 visit | Discharge through Day 15

SECONDARY OUTCOMES:
Proportion of subjects who do not receive an opioid prescription at discharge | At discharge
Proportion of subjects who do not receive a postdischarge opioid prescription, through the Day 15 visit. | Postdischarge through Day 15
Pain intensity scores at the time of discharge | At discharge
Number of oxycodone pills taken between discharge and the Day 15 visit | Postdischarge through Day 15
Mean TSQM-9 scores | Day 15 plus or minus 2 days

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Horizon Clinical Research, La Mesa, California
  - Sharp Grossmont Hospital, La Mesa, California
  - University of California, Irvine Medical Center, Orange, California
  - Parkview Community Hospital, Riverside, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Medical Research of Westchester, Inc, Miami, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - University of Louisville Hospital, Louisville, Kentucky
  - Baylor University Medical Center, Dallas, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers - New Jersey Medical School, Newark, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Hutchinson Campus, The Bronx, New York
  - M3 Emerging Medical Research, LLC, Durham, North Carolina
  - Cleveland Clinic Fairview, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - University Hospital, Columbus, Ohio
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Summit Medical Group Oregon-Bend Memorial Clinic, Bend, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - JBR Clinical Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: Undecided